CLINICAL TRIAL: NCT06679361
Title: Comparison of the Effects of Motor and Sensory Exercises on Hand Functions in Healthy Young Adults
Brief Title: Effects of Motor and Sensory Exercises on Hand Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gamze Demircioğlu, Asst. Prof. Dr., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ATLAS-MSEHF-001
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Motor Function; Retardation
Keywords: hand function; sensory; motor; exercise training; muscle reaction

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomized into three parallel groups to assess the effects of motor, sensory, and combined motor-sensory exercises on hand function. Each group will receive a specific intervention type (motor, sensory, or combined exercises), and outcomes such as muscle reaction time and hand dexterity will be measured pre- and post-intervention for both dominant and non-dominant hands.
Who Masked: Participant
Masking Description: This study will employ single masking, where participants will be unaware of their specific group assignment (motor, sensory, or combined motor-sensory exercise groups) to minimize bias. Researchers will know the group assignments to ensure correct administration of interventions, but participants will remain blinded to the type of intervention they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Motor Exercise Group (Experimental): Participants in this group will receive motor exercises targeting the wrist, including active range of motion exercises (flexion, extension, ulnar, radial deviation, and finger flexion) and nerve mobilization exercises (medial, radial, and ulnar nerves). These exercises aim to improve motor function in the wrist and hand.
  Interventions: Behavioral: Motor Exercise Program
- Sensory Exercise Group (Experimental): This group will engage in sensory exercises designed to enhance sensory awareness in the hand and wrist. Exercises will include interaction with varied textures (such as sand and sensory balls), different fabrics (fur, satin, linen), and multisensory foam gels. The goal is to improve sensory function and tactile discrimination.
  Interventions: Behavioral: Motor Exercise Program; Behavioral: Sensory Exercise Group
- Combined Motor and Sensory Exercise Group (Experimental): Arm Description: Participants in this group will perform both motor and sensory exercises as described for the first two groups. By combining motor and sensory interventions, this group aims to improve both motor skills and sensory awareness in the wrist and hand, potentially enhancing overall hand function more effectively.
  Interventions: Behavioral: Combined Motor and Sensory Exercise Group
- control (No Intervention): The control group did not receive any additional treatments during the study period, allowing for a clear comparison between the experimental group and the baseline conditions.

INTERVENTIONS:
Behavioral: Motor Exercise Program — This program consists of wrist motor exercises focused on active range of motion (including flexion, extension, ulnar and radial deviation, and finger flexion) along with nerve mobilization exercises for the medial, radial, and ulnar nerves. The aim is to enhance motor function in the wrist and hand.
  Arms: Motor Exercise Group; Sensory Exercise Group
Behavioral: Sensory Exercise Group — Arm Description: This group will engage in sensory exercises designed to enhance sensory awareness in the hand and wrist. Exercises will include interaction with varied textures (such as sand and sensory balls), different fabrics (fur, satin, linen), and multisensory foam gels. The goal is to improve sensory function and tactile discrimination.
  Arms: Sensory Exercise Group
Behavioral: Combined Motor and Sensory Exercise Group — Participants in this group will perform both motor and sensory exercises as described for the first two groups. By combining motor and sensory interventions, this group aims to improve both motor skills and sensory awareness in the wrist and hand, potentially enhancing overall hand function more effectively.
  Arms: Combined Motor and Sensory Exercise Group

SUMMARY:
This project will compare the effectiveness of sensory and motor exercises used in clinical settings for healthy young adults. This approach will allow the investigators to evaluate the impact of these exercises on hand functions.

The study plans to include 80 healthy young adults aged 18-25. After providing participants with information about the study's purpose, written informed consent will be obtained to confirm voluntary participation. Participants will be randomly assigned to one of three groups: "sensory exercise," "motor exercise," and "sensory and motor exercise." The effects on muscle reaction time and hand skills for the dominant hands will be evaluated before and after the exercises.

DETAILED DESCRIPTION:
Hand functions occupy a significant place in the functional activities of daily life. Therefore, impairments in wrist function can severely impact daily activities and quality of life. Hand rehabilitation includes various methods aimed at improving hand functions for treating numerous conditions affecting the wrist. However, it has been determined that treatments targeting both motor and sensory functions should be used together to enhance functionality. For this purpose, this project will compare the effectiveness of sensory and motor exercises used in clinical settings in healthy young adults, allowing investigators to evaluate their impact on hand functions.

The study will include 80 healthy young adults aged 18-25. After participants are informed about the study's purpose, written informed consent will be obtained to confirm voluntary participation. Participants will be randomly assigned to one of three groups: "sensory exercise," "motor exercise," and "sensory and motor exercise." The effects on muscle reaction time and hand skills for the dominant hand will be evaluated before and after the exercises. Data from the study will be analyzed using the Statistical Package for the Social Sciences (SPSS) version 25.0. Demographic characteristics of participants will be expressed as arithmetic mean ± standard deviation and percentages. The normal distribution of data will be examined using visual (histogram and probability plots) and analytical methods (Kolmogorov-Smirnov/Shapiro-Wilk tests). Pre- and post-evaluations within groups will be assessed using the student-t test, and intergroup comparisons will be evaluated with the student-t test if data follows a normal distribution, or with the Mann-Whitney U test if not. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to verbally communicate to answer questions
* Willingness to participate in the study
* Having read and signed the informed consent form

Exclusion Criteria:

* Having joint movement restriction in the upper extremity
* Presence of skin injury or scarring on the hand or wrist
* History of surgery on the upper extremity
* Having an orthopedic problem in the upper extremity
* Having a rheumatic disease
* Having a neurological condition in the upper extremity
* Having a severe mental or cognitive impairment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Hand Dexterity (Moberg Pick-Up Test) Hand Dexterity (Moberg Pick-Up Test) Hand Dexterity (Moberg Pick-Up Test) | immediately after the intervention
  This measure will evaluate hand dexterity and functional hand skills using the Moberg Pick-Up Test. Participants will be asked to place various objects into a container using both their dominant and non-dominant hands, with and without visual cues. The time taken for each attempt will be recorded, and the best score from three trials will be used to assess dexterity. Measurements are recorded in seconds, where lower scores indicate better hand dexterity.
  Scale Range: No minimum or maximum value in seconds (lower time indicates better dexterity).
  Interpretation: Lower times signify better outcomes, as they reflect quicker and more coordinated hand movements in completing the task.

SECONDARY OUTCOMES:
Muscle Reaction Time | immediately after the intervention
  Light Trainer® system, which consists of a wireless lighting system with LED pods and a central controller. The participants were seated with their hands on the table, 40 cm apart, palms down, and elbows at 90°. The Light Trainer was positioned centrally 20 cm away from each hand. When the pod was illuminated, the participants were instructed to turn off the light as quickly as possible by touching it. Light activation was randomized to avoid predictability, requiring participants to respond based on light cues each time. In the first task, the participants used their dominant hand to turn off the light as quickly as possible. In the second task, they responded to a light signal by deactivating a predetermined light from two different colors using their dominant hand.
  Scale Range: No minimum or maximum value in milliseconds (lower time is better).
  Interpretation: Lower reaction times signify better outcomes, as they reflect faster muscle response to visual stimuli.
Grip Strength (Measured Using Jamar Electronic Dynamometer) | immediately after the intervention
  Hand performance was assessed based on grip strength using a Takei Handheld Dynamometer (Takei Scientific Instruments Co., Tokyo, Japan). Participants were seated with elbows flexed at 90 degrees and forearms in a neutral position, and were instructed to squeeze the dynamometer with maximum force for 3-5 seconds, with the palm facing upwards. Each hand was tested three times with a 20-second rest between trials, and the highest value was recorded. This protocol ensures standardized and consistent results, with measurements documented in kilograms (kg) to provide reliable grip strength assessment.
  Scale Range: The dynamometer measures from 0 to 90 kg. Interpretation: Higher scores reflect stronger grip strength, which is indicative of better hand function.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study. All collected data will be used solely for the purpose of analyzing study outcomes and will remain confidential. This approach is taken to ensure the privacy and confidentiality of participant information.